CLINICAL TRIAL: NCT04569903
Title: Evaluation of a Claims-based Algorithm for the Identification of ATTR Amyloidosis in Medical Records
Brief Title: Evaluation of a Claims-based Algorithm for the Identification of Transthyretin-mediated Amyloidosis (ATTR) Amyloidosis in Medical Records
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: No patients consented to enrollment
Sponsor: Yale University (Other)
Collaborators: Alnylam Pharmaceuticals Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2000026611; 000 (Other: CTGTY)
Record Dates: First submitted 2020-09-24; First posted 2020-09-30 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Transthyretin Amyloidosis
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Computer algorithm for ATTR (Experimental): Patients will be evaluated for the identification of ATTR Amyloidosis through a claims-based algorithm
  Interventions: Device: Computer algorithm for ATTR

INTERVENTIONS:
Device: Computer algorithm for ATTR — Patients will be evaluated for the identification of ATTR Amyloidosis through a claims-based algorithm

SUMMARY:
The primary objective of this study is to evaluate the diagnostic performance of an algorithm in identifying patients with ATTR amyloidosis.

DETAILED DESCRIPTION:
A screening strategy to identify ATTR in the large background population of patients with one or more common ATTR manifestations, would be of significant clinical value.

In addition, novel ATTR therapies have been recently made available or are currently in development in late-stage clinical trials. As early diagnosis and treatment is expected to achieve better outcomes, this makes the development and validation of an easily implemented, rapid and electronically-enabled diagnostic algorithm especially important.

A medical and pharmacy claims-based algorithm was developed to potentially identify patients at risk of having ATTR. The goal of this study is to evaluate the ability of the algorithm to identify patients with ATTR by performing diagnostic clinical work up in patients that the algorithm identifies in a large dataset of patients at Yale.

The primary objective of this study is to evaluate the diagnostic performance of the algorithm in identifying patients with ATTR amyloidosis.

The secondary objective of this study is to estimate the clinical benefit of the algorithm, as measured by the added diagnostic value, i.e. the proportion or rate of patients who were previously undiagnosed. The total obtained prevalence will be assessed and informally compared to the referral-based prevalence of ATTR amyloidosis patients at Yale.

ELIGIBILITY:
Inclusion Criteria:

* Identified by the ATTR diagnostic algorithm and matched by Yale's list of potential subjects defined as:

  1. subjects within the claims dataset that are predicted to be at risk of having ATTR who are also being managed within YNHHS
  2. patients who need to be contacted and offered additional clinical evaluation to determine whether they have a diagnosis of ATTR (non-hereditary or Hereditary ATTR amyloidosis).

     Exclusion Criteria:
* Patients who have opted out of research in the Epic system will be excluded entirely from the study
* Patients who are pregnant or who may become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance of algorithm in identifying patients with ATTR amyloidosis | 2 years
  Potential thresholds for defining diagnostic positivity based on the calculated algorithmic scores will be explored and the corresponding positive predictive value (PPV) will serve as indicator for the diagnostic performance. Negative predictive values (NPV) may be explored if the actual distribution of score data will allow for it.

SECONDARY OUTCOMES:
Proportion of diagnosed patients | 2 years
  The proportion or rate of patients who were previously undiagnosed of ATTR Amyloidosis

CONTACTS AND LOCATIONS:
Overall Officials: Edward Miller, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States